CLINICAL TRIAL: NCT02358512
Title: A Phase 2 Pilot Physiological Randomised Clinical Trial to Investigate the Effect of Intermittent Versus Continuous Enteral Nutrition on Muscle Wasting in Critical Illness
Brief Title: Intermittent Versus Continuous Feeding in ICU Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University College, London (Other); The Whittington Hospital NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14\LO\1792
Record Dates: First submitted 2015-01-26; First posted 2015-02-09 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Intensive Care (ICU) Myopathy
Keywords: Intensive Care; Recovery of Function; Survivors; Outcome Assessment (Health Care); Medical Economics
MeSH Terms: conditions — Muscular Diseases | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent enteral feeding (Experimental): The intermittent feeding regimen will consist of six bolus feeds (one bolus every four hours).
  Interventions: Other: Enteral feeding
- Continuous enteral feeding (Active Comparator): The continuous feeding regimen consists of the total volume of feed administered over 24 hours.
  Interventions: Other: Enteral feeding

INTERVENTIONS:
Other: Enteral feeding — Bolus feeds or continuous feeds during a 10-day ICU stay

SUMMARY:
The purpose of this study is to determine whether intermittent nasogastric enteral feeding, rather than conventional continuous enteral feeding, will preserve muscle mass in the critically ill (Primary end-point). Such maintenance may translate into improved outcomes including reduced length of intensive care unit (ICU) and/or hospital stay, as well as number of days on a ventilator. In addition, long-term improvements in health-related quality of life and physical activity levels may result in these ICU survivors once they are back in the community. Indeed, such benefits could translate into reductions in primary healthcare usage and its related costs (secondary end-points).

DETAILED DESCRIPTION:
This is a Phase II pilot single-blinded randomized controlled trial to be conducted in two adult intensive care units. Technically, the patient will be blinded (by virtue of illness), and in any case knowledge of the feeding intervention they are receiving would not influence outcome. Scans will be taken by staff who could potentially be aware of treatment; keeping scanner personnel blinded would involve complex logistics to separate those randomising, scanning patients, and collecting data; however, the investigators don't think that the individuals taking the scans would introduce material bias. Importantly, all scans will be analysed by the same individual (based off-site) who will be blind to treatment status.

Within 24 hours of admission to ICU, patients recruited to the study will be randomised to either intermittent enteral feeding or continuous enteral feeding - both regimens delivering the same nutritional content over a 24 hour period. The intermittent feeding regimen will consist of six bolus feeds (one bolus every four hours) while the continuous feeding regimen consists of the total volume of feed administered over 24 hours. Feed volume in both groups will commence according to a standard 'usual practice' protocol so as not to delay feeding, but each patient will then have an individual regimen calculated by the dietician. Feeding will continue as either intermittent or continuous for the duration of the trial period as tolerated.

Ultrasound of the thigh (enabling derivation of the Rectus Femoris cross sectional area (RFCSA)) will be performed on Days 1,7,10 (or at discharge, if sooner), and at hospital discharge (if after Day 10), with blood and urine samples taken daily. The hospital discharge destination will be noted, and functional assessment will be determined prior to hospital discharge by two validated methods previously used in this patient cohort (6-Minute Walk Distance and Short Performance Battery Test). Patients' health-related quality of life (HRQOL) will be determined for the pre-morbid period and at 12 months post ICU-discharge using the Short Form-36 health survey; primary care costs since discharge will also be ascertained.

ELIGIBILITY:
Inclusion Criteria:

* Due to receive enteral nutrition via nasogastric tube as part of routine care; endotracheally intubated and mechanically ventilated; likely to remain intubated for 48 hours; likely to remain on the ICU for >7 days; and to survive intensive care admission.

Exclusion Criteria:

* Pregnancy
* Active disseminated malignancy (diagnosed or suspected)
* Unilateral/bilateral lower limb amputees
* Single Organ Failure (SOFA score less than 2)
* Patients with a primary neuromyopathy
* Patients entered into trials of interventions which would affect muscle mass
* Patients assessed as requiring sole/supplemental parenteral nutrition or post-pyloric feeding
* Patients requiring extra-corporeal membrane oxygenation (ECMO)
* Patients not meeting nutritional requirements in 72 hours using a standard feeding schedule
* Patients requiring the use of high protein feed
* Admission to ICU within the previous 3 months
* Ward patients who have received artificial enteral tube feeding within this hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Rectus Femoris cross-sectional area | Change between Day 1 and Day 10

SECONDARY OUTCOMES:
Length of stay on ICU | Participants will be followed for the duration of ICU stay, an expected average of 2.5 weeks
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 4.5 weeks
Discharge Location | At hospital discharge, an expected average of 4.5 weeks after admission
Number of days on ventilator | Ventilator days during ICU stay, an expected average of 2.5 weeks
6 Minute Walk Distance and Short Performance Battery Test | At hospital discharge, an expected average of 4.5 weeks after admission
  These tests will assess participant's functional ability
Health-related quality of life | 12 months post-ICU discharge
  Using Short Form-36 (SF-36) questionnaire via telephone
Number of General Practitioner (GP) and nurse consultations | 12 months post-ICU discharge
  This will provide primary care costs and allow derivation of health economic parameters, Quality-Adjusted Life Years and Cost Utility Ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hart, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Guy's & St Thomas' NHS Foundation Trust, London
  - Whittington Hospital NHS Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Puthucheary ZA, Hart N. Skeletal muscle mass and mortality - but what about functional outcome? Crit Care. 2014 Feb 17;18(1):110. doi: 10.1186/cc13729. PMID 24528611
- [Result] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Derived] Wilkinson D, Gallagher IJ, McNelly A, Bear DE, Hart N, Montgomery HE, Le Guennec A, Conte MR, Francis T, Harridge SDR, Atherton PJ, Puthucheary ZA. The metabolic effects of intermittent versus continuous feeding in critically ill patients. Sci Rep. 2023 Nov 9;13(1):19508. doi: 10.1038/s41598-023-46490-5. PMID 37945671
- [Derived] McNelly AS, Bear DE, Connolly BA, Arbane G, Allum L, Tarbhai A, Cooper JA, Hopkins PA, Wise MP, Brealey D, Rooney K, Cupitt J, Carr B, Koelfat K, Damink SO, Atherton PJ, Hart N, Montgomery HE, Puthucheary ZA. Effect of Intermittent or Continuous Feed on Muscle Wasting in Critical Illness: A Phase 2 Clinical Trial. Chest. 2020 Jul;158(1):183-194. doi: 10.1016/j.chest.2020.03.045. Epub 2020 Apr 2. PMID 32247714